CLINICAL TRIAL: NCT04518241
Title: Supporting Health Behavior Among Persons Living With HIV Using Technology, the Multiphase Optimization Strategy (MOST), and Principles of Behavioral Economics
Brief Title: Supporting Health Behavior Among Persons Living With HIV Using Tech, MOST, and Behavioral Economics
Acronym: SCAP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2020-4630
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-07

CONDITIONS: HIV Seropositivity; Adherence, Medication
Keywords: HIV; behavioral economics; adherence; HIV antiretroviral therapy; ART non-persistence; HIV non-suppression
MeSH Terms: conditions — HIV Seropositivity; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Factorial design with 3 components and 8 conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1 (Experimental): Core, fixed compensation, TMQQ, MI sessions
  Interventions: Behavioral: MI sessions; Behavioral: TMQQ; Behavioral: Type of compensation
- Condition 2 (Experimental): Core, lottery prize, TMQQ, MI sessions
  Interventions: Behavioral: MI sessions; Behavioral: TMQQ; Behavioral: Type of compensation
- Condition 3 (Experimental): Core, fixed compensation, MI sessions
  Interventions: Behavioral: MI sessions; Behavioral: Type of compensation
- Condition 4 (Experimental): Core, lottery prize, MI sessions
  Interventions: Behavioral: MI sessions; Behavioral: Type of compensation
- Condition 5 (Experimental): Core, fixed compensation, TMQQ
  Interventions: Behavioral: TMQQ; Behavioral: Type of compensation
- Condition 6 (Experimental): Core, lottery prize, TMQQ
  Interventions: Behavioral: TMQQ; Behavioral: Type of compensation
- Condition 7 (Experimental): Core, fixed compensation
  Interventions: Behavioral: Type of compensation
- Condition 8 (Experimental): Core, lottery prize
  Interventions: Behavioral: Type of compensation

INTERVENTIONS:
Behavioral: MI sessions — Three counseling sessions lasting less than 60 minutes each to identify goals, factors that promote or impede goals, and increase "readiness" for ART with high adherence
  Arms: Condition 1; Condition 2; Condition 3; Condition 4
Behavioral: TMQQ — Weekly text messages with health information as well as motivational messages. Two days later a true/false quiz question is sent. Participants earn 4 points for answering correctly, 2 points for answering incorrectly, and 0 points for not answering. Participants earn $1 for each point. Messages are sent over 21 weeks.
  Arms: Condition 1; Condition 2; Condition 5; Condition 6
Behavioral: Type of compensation — Participants who achieve HIV viral suppression at 21 weeks will receive either fixed compensation of $275 or be entered into a lottery where they have a 3/10 chance of winning $500, and a 7/10 chance of winning $175. Those who do not achieve HIV viral suppression receive a $50 participant incentive.

SUMMARY:
The present study focuses on adult persons living with HIV in the New York City and Newark, New Jersey metropolitan areas who are not highly adherent to HIV medication and who do not evidence undetectable HIV viral load (the ultimate goal of HIV treatment). Those who have not decided whether they wish to take HIV medications are invited to enroll. The study uses technology, is grounded in principles of behavioral economics, and uses the multiphase optimization strategy (MOST) to examine the acceptability, feasibility, and evidence of efficacy of three intervention components. The components are intended to increase rates of HIV viral suppression in the sample. The three components are: prizes for viral suppression (fixed compensation [$275] or lottery prizes [up to $500]), text messages and quiz questions that generate points to earn prizes (to foster engagement), and counseling sessions grounded in the motivational interviewing approach to help participants articulate goals with respect to health and viral suppression, identify and resolve barriers to HIV medication use, and build motivation for viral suppression. Participants are assessed at baseline and then 5- and 8-months later.

DETAILED DESCRIPTION:
The present study focuses on adult persons living with HIV who are not highly adherent to HIV medication and who do not evidence undetectable HIV viral load (the ultimate goal of HIV treatment). The study uses technology, is grounded in principles of behavioral economics, and uses the multiphase optimization strategy (MOST) to examine the acceptability, feasibility, and evidence of efficacy of three intervention components. The components are intended to increase rates of HIV viral suppression in the sample. All participants receive a core intervention comprised of referrals to care and case management. The three components are: compensation for viral suppression (fixed compensation or lottery-type prizes), weekly text messages and quiz questions (TMQQ) for 21 weeks that generate points to earn compensation (to foster engagement), and three counseling sessions grounded in the motivational interviewing (MI) approach to help participants articulate goals with respect to health and viral suppression, identify and resolve barriers to HIV medication use, and build motivation for viral suppression. We have previously tested variations of these components together as a "packaged" intervention and found high acceptability, feasibility, and evidence of efficacy. We now seek to understand this approach with more precision by testing the effects of individual components using MOST. The components will be tested in a factorial design with 8 intervention conditions. Consistent with the factorial design, each condition will comprise a unique combination of components. Each condition includes at least one component. Participants will be recruited by a proven hybrid strategy that includes peer recruitment, ads placed in a free newspaper, and direct recruitment from an NYU Recruitment Registry managed by Dr. Gwadz. Participants will be screened for eligibility and a total of 80 adult persons living with HIV and with detectable HIV viral load will be enrolled in the study and randomly assigned to an intervention condition. Participants will be assessed at baseline and 5- and 8-months post-baseline with a structured assessment battery. A subset will receive in-depth interviews. The primary outcome is viral suppression. This is a pilot study. It is not powered for efficacy but we will examine evidence of efficacy. All study activities can be carried out in a virtual format, and we can switch to in-person contact for screening, assessment, and some components when appropriate. In-person activities would be conducted at the New York University Silver field site in Manhattan. The study is funded through the Constance and Martin Silver Artificial Intelligence and Social Impact Fund at the New York University Silver School of Social Work.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Has diagnosis of HIV infection
* Resides in the New York City or Newark, NJ metropolitan areas
* Can conduct research activities in English
* Has a phone that can send and receive text messages
* Has not participated in a conditional economic incentive program for HIV viral suppression in the past month
* Has not been enrolled in this research team's two recent studies
* Has detectable HIV viral load (> 200 pp/mL) by lab report

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Undetectable HIV viral load | 5-months post-baseline
  achievement of undetectable HIV viral load (< 200 pp/mL)
Undetectable HIV viral load | 8-months post-baseline
  achievement of undetectable HIV viral load (< 200 pp/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Marya Gwadz, PhD, Principal Investigator — New York U
Locations (1):
- New York University Silver School of Social Work, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Filippone P, Serrano S, Gwadz M, Cleland CM, Freeman R, Linnemayr S, Cluesman SR, Campos S, Rosmarin-DeStefano C, Amos B, Israel K. A virtual pilot optimization trial for African American/Black and Latino persons with non-suppressed HIV viral load grounded in motivational interviewing and behavioral economics. Front Public Health. 2023 May 10;11:1167104. doi: 10.3389/fpubh.2023.1167104. eCollection 2023. PMID 37234760